CLINICAL TRIAL: NCT07093489
Title: Evaluation of the Effectiveness and Safety of the LC16m8 Mpox Vaccine in Individuals Aged One Year and Older in the Democratic Republic of Congo (DRC)
Brief Title: Evaluation of Effectiveness and Safety of LC16m8 Mpox Vaccine in the Democratic Republic of Congo (DRC)
Acronym: MPX-001
Status: Not yet recruiting | Type: Observational
Sponsor: International Vaccine Institute (Other)
Collaborators: Japan Institute for Health Security (JIHS) (Unknown); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Other Study IDs: MPX-001
Record Dates: First submitted 2025-07-07; First posted 2025-07-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mpox (Monkeypox); Mpox
Keywords: LC16m8; Mpox; Effectiveness; Safety; DRC
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox vaccine LC16m8

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples With DNA — Skin swabs will be collected from all patients presenting with skin lesions suggestive of mpox. Oro-pharyngeal swabs and saliva will be collected from one hundred Consecutively invited patients with skin lesions to assess the diagnostic accuracy of other samples compared to skin swab. In patients without skin lesions, oro-pharyngeal swab will be collected. Skin lesion material includes swabs of lesion surface and/or exudate, or lesion crusts. Lesions will be swabbed vigorously to ensure adequate viral DNA is collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort Event Monitoring (CEM) - Safety cohort: At enrollment/vaccination visit, participants will be consecutively invited to be enrolled in the safety subset until the sample size of 10,000 has been achieved. The enrollment aims to include a proportional number of participants from various age groups, including 1-5 years, 6-12 years and 13-18 years, with representation from both sexes. The participation will be strictly voluntary according to the eligibility criteria.
  Enrolled vaccinees will be actively followed up through phone calls/home visits/Health facility visits for the SAEs and AESIs assessment at weekly intervals for the first month and then at monthly intervals until 12 weeks post vaccination. Vaccinees/parents/guardians will be advised to return to the sentinel health facility if any serious event occurs at any time.
  Interventions: Biological: LC16m8
- Vaccine Effectiveness (VE) Assessment: Health facility-based enhanced mpox surveillance will be implemented to record mpox cases within the vaccination catchment area. The study will be done in 2 or more health zones identified as hot spots by the DRC government. All patients presenting with probable or suspected mpox to the surveillance healthcare facilities will be approached for testing and enrollment into the surveillance study.
  Vaccine effectiveness will be estimated using cases and controls assembled based on specific inclusion/exclusion criteria. A total of 1,990 participants (398 cases and 1,592 controls) will be required for assessment of vaccine effectiveness.

INTERVENTIONS:
Biological: LC16m8 — LC16m8 vaccine will be offered to all individuals aged >1 year and meet the inclusion criteria within the catchment population. This will be done in line with the DRC government's LC16m8 vaccine roll out plan.
  Groups: Cohort Event Monitoring (CEM) - Safety cohort

SUMMARY:
This is a health facility-based prospective test-negative (TND) case-control study to evaluate vaccine effectiveness and active safety monitoring (cohort event monitoring), and passive surveillance for evaluation of the safety of the LC16m8 mpox vaccine in individuals aged one year and older in the DRC.

This study aims to assess the LC16m8 vaccine effectiveness and safety. The following activities will be carried out:

* Community engagement
* Enhanced health facility-based mpox disease surveillance
* Vaccination using the LC16m8 vaccine
* Safety monitoring following immunization
* LC16m8 Vaccine effectiveness evaluation using a TND

Study Hypothesis: The LC16m8 vaccine, administered as pre-exposure prophylaxis, confers greater than 70% protection against symptomatic mpox disease among adults and children in the DRC.

DETAILED DESCRIPTION:
1. Community Engagement: The community mobilization will be carried out according to the national communication plan for the vaccination promotion. Study staff members will engage with religious leaders, medical professionals, heads of villages, and key opinion leaders to share information about the mpox disease surveillance, the availability of the vaccine, and the vaccination. Additionally, detailed information regarding the available mpox testing and treatment facilities that the community needs to visit if any person develops symptoms consistent with mpox or develops adverse events following vaccination will be provided in the community engagement activities. Special emphasis will be made in the community messaging to encourage all individuals with mpox-compatible symptoms regardless of the disease severity and vaccination status-to promptly seek testing and care.
2. Enhanced Health Facility-based Mpox Disease Surveillance: Health facility-based and enhanced mpox surveillance will be implemented to record mpox cases within the vaccination catchment area. The study will be done in 2 or more health zones identified as hot spots by the DRC government.

   The healthcare facilities within the study catchment area will be equipped with mpox testing equipment & supplies and the study staff will receive comprehensive training for the mpox case investigation, sample collection, and management. Pre-existing laboratories will be supported by the project to perform RT-PCR tests, and a subset of samples will be shipped to the reference microbiology laboratory at INRB headquarters in Kinshasa for quality control.

   Patients presenting at a sentinel surveillance healthcare facility with suspected or probable mpox will be approached for enrollment. For patients presenting with skin lesions, a swab of the skin will be collected from all suspected/probable mpox cases for testing using RT-PCR. Out of the patients presenting with skin lesions, one hundred patients will be consecutively invited to provide oro-pharyngeal swab and saliva to assess the diagnostic accuracy of other samples compared to skin swab. For patients presenting without skin lesions, oro-pharyngeal swab will be taken. Each suspected case will be asked for contact information (telephone number and/or description of residence). After 3 weeks, study staff will seek to contact, by telephone and/or in-person visit, each suspected case who tested negative by RT-PCR at enrollment to assess whether or not the individual experienced additional symptoms and signs consistent with symptomatic mpox, particularly the development of skin lesions. The study staff will seek to collect skin or oropharyngeal swabs from initially test-negative patients who reported experiencing additional symptoms consistent with symptomatic mpox during the three-week period after enrollment and to test these samples by RT-PCR.
   1. Laboratory Procedure: Real-time polymerase chain reaction (RT-PCR) for the presence of MPXV in skin swabs from all patients presenting with skin lesions suggestive of mpox will be performed for laboratory confirmation and diagnosis of mpox. For patients presenting without skin lesions, oro-pharyngeal swab will be tested using RT-PCR. The RT-PCR protocols for the detection of MPXV will be performed according to manufacturer's instructions, in line with WHO guidelines for the detection of MPXV.
   2. Specimen Type, Collection, Transport and Storage: Skin lesion material includes swabs of lesion surface and/or exudate, or lesion crusts. Lesions will be swabbed vigorously to ensure adequate viral DNA is collected. Swabs will either be transported dry in capped tubes or placed in viral transport media (VTM). Whenever possible, specimens from two lesions should be collected in one single tube, preferably from different locations on the body. For patients with no skin lesions at presentation, oro-pharyngeal swabs will be taken. Samples will be stored at 2-8°C if processed within 72 hours. Samples that are shipped to reference laboratories will be stored at -20°C or lower. Longer-term storage (>60 days) will be at -70°C. All specimens being transported should have appropriate triple packaging, labelling, and documentation.
3. Vaccination using LC16m8 Vaccine: As the study aims to generate real-world vaccine effectiveness by leveraging DRC's national mpox vaccination strategy, the vaccination will be conducted in 2 to 3 selected health zones/areas which meet the criteria for a hotspot as defined by the DRC vaccination strategy for targeted vaccine delivery.

   Selection of health zones/area for the study where LC16m8 is expected to be offered to everyone one year or older, will be determined based on the latest mpox epidemiological data, operational feasibility, and existing research infrastructure in close consultation with DRC MoH, Institut National de Santé Publique (INSP), and local stakeholders. Due to on-going mpox outbreaks in multiple provinces in DRC, investigators will also ensure enough doses are allocated and delivered to selected health zones/areas to reach minimum coverage required for the study (i.e., 30% coverage). Details of the vaccination strategy will be determined in close collaboration with local public health authorities.

   a. Vaccination Information Registration: As mpox vaccine is being offered as part of DRC's national mpox vaccination strategy, consent/assent procedure for the vaccination will be carried out according to the routine public health immunization program. Vaccination sites/centers will collect mpox vaccination registry as per routine practice as well and provide a vaccination card along with detailed instructions on how to securely retain it for future reference.

   In addition to routine immunization practices, each person receiving LC16m8 vaccine in selected health zones/areas will be asked to provide biometric information (i.e., iris scanner). Study staff will collect informed consent/assent from vaccinees prior to collecting any biometric data. Collected biometric information along with mpox immunization records will be registered to a dedicated database (e.g., REDCap platform), which will be maintained by the INRB. In case vaccinees reject to provide any biometric information for the study purpose, only paper-based immunization registry will be collected as per routine practice.

   For those who agreed to provide biometric information, vaccination records will be merged with provided biometric information. For paper-based registry, it will be entered into electronic vaccination database (i.e., REDCap platform managed by INRB). The vaccination database will include key personal identifiers, which will be used in an electronic "parsing tool," such as the one developed in-house by the International Vaccine Institute (IVI), which is a software capable of linking sociodemographic data of an individual to a vaccine registry database. Biometric information and/or "parsing tool" on electronic vaccination database will be used to correctly identify mpox vaccination history for those enrolled into the test-negative case-control study to enable calculation of VE estimates
4. Safety Monitoring Following Immunization with LC16m8 Vaccine: All participants receiving the LC16m8 vaccine will be observed for the first 30 minutes of vaccination as per the DRC's national vaccination strategy. The monitoring of the LC16m8 vaccine safety administered during vaccination will be assessed through:

   1. A cohort event monitoring (CEM), an observational prospective cohort study: At enrollment/vaccination visit, participants will be consecutively invited to be enrolled in the safety subset until the sample size of 10,000 has been achieved. The enrollment aims to include a proportional number of participants from various age groups, including 1-5 years, 6-12 years and 13-17 years, with representation from both sexes. Enrolled vaccinees will be actively followed up through phone calls/home visits/Health facility visits for the SAEs and AESIs assessment at weekly intervals for the first month and then at monthly intervals until 12 weeks post vaccination. Vaccinees/parents/guardians will be advised to return to the sentinel health facility if any serious event occurs at any time. All adverse events including AESIs and SAEs will be assessed using CRFs adapted from existing tools from WHO protocol. All SAEs and AESIs will be assessed for relatedness, seriousness, expectedness, and outcome.

      Participants will have the right to withdraw from the study at any time and for any reason. Withdrawn participants will not be replaced after the recruitment of participants has ended. Data collected from withdrawn participants will be used for study purposes. A participant will be considered as lost-to follow-up after three documented unsuccessful attempts have been made to contact the participant, by phone/home visit. Participants that are lost to follow-up will not be replaced after the enrollment is completed.
   2. A passive surveillance at sentinel surveillance sites: Passive AEFI surveillance will be conducted at designated health facilities within the catchment area. Therefore, data on SAEs & AESI will be collected through health facility records or voluntarily reporting of event(s) by the vaccinees/parents or guardians (self-reported data) and by healthcare workers. Medical records in these facilities will be regularly reviewed to detect any potential serious adverse events or AESIs associated with vaccination including adjudication of causality, relatedness, seriousness and temporal relationship with vaccination. Potential SAEs and AESI will be recorded in dedicated forms by a trained health professional. Vaccination data will be linked to the passive surveillance data using the same database/parsing tool used for vaccination ascertainment in the VE study.

   Female study participants of childbearing age will be instructed to report to the study staff any pregnancy case which occurs within three months after receiving the vaccine. Pregnant women who are inadvertently exposed to the LC16m8 vaccine and women who become pregnant within 3 months of vaccination will be followed every three months until delivery or the end of pregnancy. The neonatal and maternal outcomes will be recorded based on records at the health facility. Pregnancy itself is not considered an AEFI, but any complications during pregnancy are to be considered as AEFI, and in some cases could be considered Serious AEFI. Spontaneous abortions, blighted ovum, fetal death, stillbirth, an elective termination for medical rationale and congenital anomalies reported in the baby are always considered as Serious AEFI, and the information should be provided using an appropriate Serious AEFI form.

   SAE and AESIs will be actively monitored over 12 weeks after immunization in the safety cohort and throughout the study duration as part of passive surveillance.
5. LC16m8 Vaccine Effectiveness using the Test-Negative Design: An observational, prospective, health facility-based study, following the TND will be carried out in each participating site to assess the effectiveness of vaccination using the LC16m8 vaccine. In the TND study, the cases and controls are both seeking services for mpox diagnostic testing and management because of mpox-like illnesses - the cases being those testing positive for mpox using RT-PCR and the controls those testing negative . As such, the bias introduced by healthcare-seeking differences is controlled by implementing TND study for vaccine effectiveness (VE) evaluation by disease severity.
6. Statistical Considerations

   1. Sample Size

      * Sample Size for the VE Assessment: Vaccine effectiveness will be estimated using cases and controls assembled based on specific inclusion/exclusion and matching criteria. Detailed matching procedures will be described in the statistical analysis plan (SAP). Assuming a vaccine effectiveness of 70%, 20% precision, 30% vaccine coverage among the controls, response rate of 80%, and a case-to-control ratio of up to 1:4, a total of 1,990 participants (398 cases and 1,592 controls) will be required to estimate VE.
      * Sample Size for the Safety Assessment: Assuming that at least one event with an event frequency of 1 per 3,333 will be observed with 95% CI, the required sample size for the CEM will be 10,000 stratified by age group.
   2. Statistical Analysis: For statistical analysis, there will be two data sets: safety data set which will be used for analysis of safety and surveillance data set which will be used for analysis of vaccine effectiveness. The details of the statistical considerations for each of the endpoints will be addressed in the dedicated SAP. This section presents the high-level summary of the analysis considerations.

      * Analysis of Safety Data: The analysis of SAEs and AESIs will include data for all participants. Participation rates over time will be described. Demographic characteristics will be summarized. In addition, descriptive analysis will be done on subgroups of different age strata. Information on baseline characteristics and potential covariates such as: medical history and concomitant medicines will be collected.

   Observed-to-expected analyses will be performed for SAEs and AESIs with an unknown risk window. The observed incidences for AESIs will be compared with background rates from the most appropriate sources including good quality national background rates will be used if available. Sensitivity analyses will be performed if deemed appropriate. The expected rate will be age and sex-stratified, and the standardized incidence ratio (SIR) will be calculated. In addition, the frequency and proportion of participants with at least one SAE or AESI will be calculated overall, by event type and by time since receipt of mpox vaccine, in days. For each type of event, the duration (in days) will be calculated, and their mean/median and standard deviation/range will be reported as well as any sequelae. A cumulative incidence will be calculated and plotted to visualize trends and identify inconsistent/unexpected patterns. For acute AESIs with a known risk window, a self-controlled risk interval analysis will be considered provided the risk window for the adverse event of interest is within 42 days, to allow sufficient time for the control period. For the proportions, the 95% confidence intervals will be calculated using an exact method. For each type of event and severity, the duration (in days) will be calculated, and their mean/median and standard deviation/range will be reported.

   • Analysis of Vaccine Effectiveness: The primary test-negative evaluation will define cases as those who test positive by RT- PCR for mpox at enrollment, and controls will be selected for inclusion from among those who were RT-PCR-negative at enrollment. To adjust for potential bias related to the selection of controls, additional test negative evaluations including based on testing (at enrollment and at three weeks follow up) of those without a skin lesion at presentation will be performed. Additionally, vaccinated and unvaccinated test negative controls will be compared for the incidence of non-vaccine targeted infections such as varicella . Details of these analyses will be presented in the SAP. Selection of cases and test-negative controls for all test-design analyses will be conducted by an individual who will not have access to information about the LC16m8 status of these individuals.

   For the primary endpoint analysis (VE against RT-PCR confirmed mpox), the investigators will use conditional multivariable logistic regression analysis to adjust for confounding variables. Health zone, age, sex, calendar date of testing, mpox severity at presentation, Charlson Comorbidity Index, and history of smallpox vaccination or disease, and others as appropriate will be considered as confounders, the final VE estimates will be calculated using the adjusted odds ratio (aOR) for vaccination using the following formula: VE = (1-aOR) × 100%. Imputation of missing values in the data will be considered based on the level of missing data and the distribution of the data. The procedures for imputation will be described in the SAP. The investigators will quantify and measure the precision of any effect modification or confounding including for VE estimation by subgroup. If effect modification exists, VE and CIs will be reported for each subgroup separately. Odds ratios will be estimated by exponentiation of the coefficient for vaccination in the models, and standard errors for these coefficients will be used to calculate 2-sided p-values and 95% confidence intervals for the ORs for TND. VE for the primary endpoint will be calculated separately for different vaccination status, complete vaccination, incomplete vaccination and unvaccinated. The investigators will evaluate the goodness of fit, identification of outliers, and the presence of multiple co-linearity.

   Using the propensity score, the investigators will calculate the inverse probability of receiving the LC16m8 mpox vaccine weighting. The propensity score will be estimated using the Generalized Boosted Regression Models (GBM) approach based on age, sex, calendar date of testing, mpox severity at presentation, Charlson Comorbidity Index, and history of smallpox vaccination or disease. The investigators will conduct the weighted logistic regression analysis using inverse probability weighting to estimate VE and its 95% confidence interval.
7. Data Management: Data management will be coordinated by INRB and will be supported by IVI using validated databases (example, REDCap). All the data generated during the conduct of the study will be entered into the paper Case Report Form (CRF) and will be transcribed in respective electronic Case Report Forms (eCRF) or directly entered onto the eCRF for each participant enrolled in the study.

Study staff will extract all data collected in source documents and workbooks for computerization into the eCRF when required. Data will be entered into computers in a dedicated area located using data entry programs specially created for the study. All programs will incorporate identification of the key punching errors, range, and consistency checks with data entry. This data management system will provide error reports and summary reports for each activity. The database management system will be guided by the principles that govern biomedical research involving human subjects, the Declaration of Helsinki, and Good Clinical Practice (GCP). It will ensure participant confidentiality by not allowing users to link names with the history of medical events of the study participants. Access to the electronic database and hard-copy data will be restricted to authorized study personnel only. The data will be automatically backed up systematically onto study site or IVI or representative server. In addition, the software will provide an audit trail of all sequential changes made. Data security will be augmented by automatic computer virus scanning at start-up of data entry and data management session, and password protection for accessing data and data management software. Data entry and cleaning will be conducted at the sites. Final data cleaning, data freezing, and data analysis will be performed by IVI or designated implementing partners. All data documents, including systems documents, forms, error outputs and resolutions, will be kept in a locked file cabinet for future reference. Necessary measures will be taken so that forms are protected from hazards such as rot, insects, and theft. Since a database could be damaged or lost in many ways, backup files will be kept, and backups will be made regularly onto external storage devices. Multiple backups of at least the last three generations (an update in the database creates a new generation of database) of the database will be kept since errors found in a recent data set might require reviewing a previous copy of it. One backup copy will be kept in a geographically separate location. The logs of every backup will be maintained in a logbook that contains the database name, name of the person who conducted the backup, backup date, media name, and location of the media.

ELIGIBILITY:
1. Vaccination:

   Inclusion criteria
   * Individuals aged 12 months and above
   * Living in the study catchment area
   * Written informed consent/assent (if applicable)

   Exclusion criteria
   * Prior receipt of any mpox vaccine dose
   * Women known to be pregnant or breast feeding
   * Individuals suffering from any spreading skin disease
   * Immunocompromised individuals with known severe immuno-deficiency conditions (example, HIVAIDS, individuals being on chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisolone equivalent for periods exceeding 10 days, cytotoxic or other immunosuppressive drugs)
   * Individuals with known underlying uncontrolled chronic diseases such as diabetes mellitus, cardiovascular disease, renal disease, hepatic disease, hematological disease, and developmental disturbance
   * Individuals with a history of hypersensitivity caused by a component of the vaccine

   Temporary exclusion criteria
   * Individuals with objective fever (Frontal temperature ≥ 38.5°C) or axillary temperature > 37.5 °C
   * Individuals suffering from acute illness within 48 hours prior to vaccination and based on investigator judgement.
   * Receipt of any live vaccine injection within the previous 27 days (measles vaccine, rubella vaccine, mumps vaccine, varicella vaccine, BCG vaccine, yellow fever vaccine...).
2. Cohort Event Monitoring (CEM):

   Inclusion criteria
   * Written informed consent
   * Individual who receives single dose of LC16m8 vaccine at one of the vaccination centers participating in the study.
   * Must be reachable by phone (must have an active phone number of his/her own or in the household) throughout study participation.

   Exclusion criteria

   • Individual/parent/guardian unable to comply with the study procedures
3. Mpox surveillance (VE):

General Inclusion Criteria:

* Patients (with any vaccination status) presenting to a sentinel surveillance health facility with clinical signs and symptoms consistent with mpox disease (probable or suspected)
* Reside in the study area prior to testing.
* Eligible to receive LC16m8 vaccine during the vaccination.
* Give consent/assent (if applicable) to participate in the study.

Exclusion Criteria

* Individuals meeting any of the following criteria are not eligible for testing and enrollment in the study:
* Known contraindications for LC16m8 vaccine.
* As per the Investigator's medical judgement, an individual could be excluded from the study despite meeting all the inclusion/exclusion criteria mentioned above.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The vaccination will be conducted in 2 to 3 selected health zones/areas which meet the criteria for a hotspot as defined by the DRC vaccination strategy for targeted vaccine delivery. As of February 2025, the DRC government has updated their comprehensive mpox vaccination plan which targets both high-risk groups (e.g., healthcare workers, contacts of confirmed cases, etc.) as well as population residing in 57 health zones considered mpox hotspots based on recent epidemiologic data.
  Selection of health zones/area for the study, where LC16m8 is expected to be offered to everyone one year or older, will be determined based on the latest mpox epidemiological data, operational feasibility, and existing research infrastructure in close consultation with DRC MoH, Institut National de Santé Publique (INSP), and local stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 11990 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with complete mpox vaccination among those with symptomatic, RT-PCR confirmed mpox infection compared to those who test negative for mpox RT-PCR. | At baseline (Day 0)
  This outcome measures the percentage of participants who had complete vaccination among those who tested positive for mpox by RT-PCR in comparison to the percentage of participants who had complete vaccination who tested negative for mpox by RT-PCR.
  Unit of Measure: Odds ratio
  Measurement tool: The odds of complete Vaccination status determined through vaccination record or participant self-report (complete vaccination is defined as symptom onset ≥14 days after receiving mpox vaccine) among mpox positive cases (RT-PCR positive) compared to the odds of complete Vaccination status among controls (mpox RT-PCR negative).

SECONDARY OUTCOMES:
The percentage of participants with complete vaccination in different age strata of participants with RT-PCR-confirmed mpox disease compared with the percentage of participants with complete vaccination in those without mpox disease. | At baseline (Day 0)
  This outcome will assess the correlation between mpox disease status and vaccination status at the time of enrollment. Specifically, the investigators will compare the odds of having received a complete mpox vaccination among participants with RT-PCR-confirmed mpox disease to the odds among those who test negative for mpox. Analyses will be stratified by age group to explore potential age-related differences in vaccine coverage and effectiveness. Complete vaccination is defined as onset of first mpox symptoms 14 days or more after receipt of mpox vaccine.
  Unit of measure: Odds ratio
  Measurement tool: The odds of complete vaccination status (complete vaccination is defined as symptom onset ≥14 days after receiving mpox vaccine) in among mpox positive cases (RT-PCR positive) compared to the odds of complete Vaccination status among controls (mpox RT-PCR negative).
The percentage of participants with incomplete vaccination among participants with RT-PCR-confirmed mpox disease compared to the percentage of participants with incomplete vaccination among participants with negative mpox RT-PCR(overall&stratified by age | At baseline (Day 0)
  This outcome measures the odds of having an incomplete mpox vaccination status among participants with RT-PCR-confirmed mpox at the time of enrollment compared to participants who test negative to mpox. Incomplete vaccination is defined as onset of first mpox symptoms within 14 days of receipt of mpox vaccine. The analysis will be conducted both overall and stratified by age to examine potential differences across age groups.
  Unit of measurement: Odds ratio
  Measurement tool: The odds of incomplete vaccination status (incomplete vaccination is defined as symptom onset within 14 days of receiving mpox vaccine) among mpox positive cases (RT-PCR positive) compared to the odds of incomplete Vaccination status among controls (mpox RT-PCR negative).
The percentage of participants with complete vaccination in those with RT-PCR-confirmed severe mpox disease compared to the percentage of participants with complete vaccination in those without mpox (overall & stratified by age). | From baseline (Day 0) to severe outcome (death or hospitalization, assessed up to Day 42)
  This outcome assesses whether complete vaccination is associated with reduced odds of developing severe mpox disease. Odds of complete vaccination will be compared between participants with RT-PCR-confirmed severe mpox and those without mpox, both overall and stratified by age. Complete vaccination is defined as onset of first mpox symptoms 14 days or more after receipt of mpox vaccine.
  Unit of measurement: Odds ratio
  Measurement tool: The odds of complete Vaccination status (complete vaccination is defined as symptom onset ≥14 days after receiving mpox vaccine) among mpox positive cases (RT-PCR positive) compared to the odds of complete Vaccination status among controls (mpox RT-PCR negative).
The percentage of participants with incomplete vaccination in those with RT-PCR-confirmed severe mpox disease compared to the percentage of incomplete vaccination among those without mpox disease (overall & stratified by age). | From enrollment (Day 0) to severe outcome (death or hospitalization, assessed up to Day 42)
  Comparison of the odds of incomplete vaccination status between participants diagnosed with RT-PCR-confirmed severe mpox disease and those without mpox disease, overall and stratified by age groups. Incomplete vaccination is defined as onset of first mpox symptoms within 14 days of receipt of mpox vaccine.
  Unit of measurement: Odds ratio
  Measurement tool: The odds of incomplete vaccination status (incomplete vaccination is defined as symptom onset within14 days of receiving mpox vaccine) among mpox positive cases (RT-PCR positive) compared to the odds of incomplete vaccination status among controls (mpox RT-PCR negative).
Evaluate the incidence of serious adverse events (SAEs) and adverse event of special interest (AESI) of the LC16m8 vaccine using a cohort event monitoring (CEM) in a defined cohort and passive surveillance in all vaccinees. | Within 12 weeks following immunization in the CEM cohort and with 12 months in the rest of the vaccinees (not part of the CEM cohort)
  Monitor and assess the occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) following administration of the LC16m8 vaccine through active cohort event monitoring (CEM) in a specified group and passive surveillance in all other vaccine recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Jacques Muyembe, Principal Investigator — Institut National de la Recherche Biomédicale; Norio Ohmagari, Principal Investigator — Japan Institute for Health Security; Florian Marks, Study Chair — International Vaccine Institute
Locations (1):
- The Institut National de la Recherche Biomédicale (INRB), Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No